CLINICAL TRIAL: NCT01165385
Title: An Open Label Dose Escalation and Pharmacokinetic Phase I Study With Pazopanib in Combination With Cisplatin (CDDP) Every Three Weeks in Patients With Advanced Solid Tumors
Brief Title: Study With Pazopanib in Combination With Cisplatin (CDDP) in Patients With Advanced Solid Tumors
Acronym: PACIFIK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEP 07/0908 - PACIFIK
Record Dates: First submitted 2010-06-25; First posted 2010-07-19 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Solid Tumors; Metastatic Cancer
Keywords: Relapsed or refractory solid tumors; Pazopanib; Cisplatin
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence | interventions — Cisplatin; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib and Cisplatin (Experimental): * Steady state period:Pazopanib will be given 8 days prior to cisplatin
  * Then pazopanib will be given 400 mg, 600 mg or 800 mg/day, daily and cisplatin 60, 75 or 100 mg/m2 , day 1 - 3 weekly, depending of the dose level
  Interventions: Drug: cisplatin; Drug: Pazopanib

INTERVENTIONS:
Drug: cisplatin — 60, 75 or 100 mg/m2 , day 1 - 3 weekly
  Other Names: Cisplatinum
Drug: Pazopanib — 400 mg, 600 mg or 800 mg/day, daily
  Other Names: GW76034

SUMMARY:
The aim of this research is to evaluate the potential interest of an association of Pazopanib, a multi-tyrosine kinase inhibitor, and cisplatin.

As cisplatin has marketing approval for several cancers (ovarian, testicle, bladder, esophagus, endometrium, lung, stomach, head and neck cancer (HNC)), and in order to have a rapid evaluation of this combination, we will evaluate the combination in any patient whose tumors is known to be sensible to cisplatin (except tumors at risk of bleeding).

This study is a classical phase 1 trial of pazopanib and 3-weekly cisplatin association. It will allow for optimal dose selection and pharmacokinetic analysis. It is planed to include around 38 patients, enriching the optimal tolerated regimen (OTR) level only with a cohort of triple negative breast cancer patients. If the association is proven to be feasible, we will then move to a specific phase II study in triple negative breast cancer patients.

DETAILED DESCRIPTION:
The main objective of the study is to determine the dose limiting toxicities (DLT) and the optimal tolerated regimen (OTR) which are both safety criteria evaluated upon the NCI CTC-AE system version 4.0.

Efficacy is not the primary objective; however the anti-tumor activity of the pazopanib/cisplatin combination will be carried out by the determination of the objective response rate according to RECIST criteria version 1.1.

The objective response is defined as either a complete response (CR) or partial response (PR), assessed either by CT Scan and/or MRI and/or bone Scan, performed at baseline and every 6 weeks.

This is an open-label, non-randomized, dose escalation and pharmacokinetic, phase I study pazopanib with cisplatin in patients with relapsed or refractory solid tumors (except tumors at risk of bleeding) for whom the selected combined chemotherapy is indicated or is a reasonable option (as per tumor characteristics and previous treatments).

All eligible patients entering the study will receive daily oral pazopanib, supplied as 200 mg aqueous film-coated tablets and intravenous cisplatin every three weeks. Doses of both compounds will be adjusted according to the reached dose level.

The treatment will continue until the development of unacceptable toxicity or evidence of disease progression or until patient's / investigator's decision of withdrawal.

All patients who received at least on dose of the study drug will be followed for survival outcome.

ELIGIBILITY:
Main Inclusion Criteria:

* Documented metastatic solid malignancies for patients who are candidate to receive a cisplatin based regimen.

  * During the dose seeking procedure : ALL solid tumors
  * During the Optimal Tolerated Regimen validation procedure : ONLY HER2-RH- breast cancer
* Measurable or evaluable disease
* WHO performance status ≤ 1
* Negative dipstick proteinuria test or if positive proteinuria <1g/24h. If proteinuria appears ≥ 2+ on routine dipstick testing, patients must undergo a 24H -urine collection and demonstrate proteinuria < 1g/24H
* Corrected QT interval (QTc) ≤ 480 msecs using Bazett's formula

Main Exclusion Criteria:

* Prior treatment with cisplatin reaching a cumulative dose> 300 mg/m2
* HER2 positive breast cancer
* Patients at high risk of bleeding
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
* calcium and magnesium levels inferior to standard levels (measured within 14 days before the first pazopanib dose) and potassium levels inferior to standard levels (measured within 72 hours before the first pazopanib dose)
* Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study
* Hearing impairment/tinnitus > or = grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Determination of the Optimal Tolerated Regimen (OTR) based on the occurrence of Dose Limiting Toxicities | cycles 1 and 2

SECONDARY OUTCOMES:
Objective response - Overall Objective response rate - Clinical Benefit Rate | At baseline and every 6 weeks.
  Anti-tumor activity of the pazopanib/cisplatin combination will be carried out by the determination of the objective response rate according to RECIST criteria version 1.1.
To characterize the pharmacokinetic (PK) profile of the combination pazopanib and cisplatin | Cycles 1 and 2
  The objective of the pharmacokinetics is to investigate the interactions between cisplatin IV and pazopanib

CONTACTS AND LOCATIONS:
Overall Officials: Veronique DIERAS, MD, Study Chair — Institut Curie
Locations (5):
- France (5):
  - Centre François BACLESSE, Caen
  - Centre Georges François LECLERC, Dijon
  - Centre Léon Berard, Lyon
  - Centre René Gauducheau, Nantes Saint Herblain
  - Institut Curie, Paris

REFERENCES:
- [Derived] Dieras V, Bachelot T, Campone M, Isambert N, Joly F, Le Tourneau C, Cassier P, Bompas E, Fumoleau P, Noal S, Orsini C, Jimenez M, Imbs DC, Chatelut E. A Phase I, Dose-Escalation Trial of Pazopanib in Combination with Cisplatin in Patients with Advanced Solid Tumors: A UNICANCER Study. Oncol Ther. 2016;4(2):211-223. doi: 10.1007/s40487-016-0027-x. Epub 2016 Aug 18. PMID 28261651